CLINICAL TRIAL: NCT02736136
Title: An Early Intervention to Increase Maternal Self-efficacy After Preterm Birth
Acronym: JOIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Antje Horsch, Research psychologist, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 496/15
Record Dates: First submitted 2016-04-04; First posted 2016-04-13 (Estimated); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Posttraumatic Stress Disorder; Stress; Anxiety; Depression
Keywords: maternal parenting self-efficacy; parental stress; maternal sensitivity; mother-infant bond
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Joint observation and video feedback plus usual care in the neonatology (plus completion of self-report questionnaires and 15 min filmed mother-infant interaction)
  Interventions: Behavioral: joint observation and video feedback
- Control (No Intervention): Usual care in the neonatology (plus completion of self-report questionnaires and 15 min filmed mother-infant interaction)

INTERVENTIONS:
Behavioral: joint observation and video feedback
  Arms: Intervention

SUMMARY:
This study aims to investigate the effects of an early intervention (joint observation and video feedback) on maternal parenting self-efficacy following a premature birth. Mothers who have given birth to a very premature baby will be randomly allocated to either the early intervention or usual care whilst the infant is still hospitalized. Participants will be followed up at one month and six months. It is predicted that participants who received the early intervention will report higher maternal parenting self-efficacy than those who are not.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of very preterm infants born between 28 and 32 weeks of gestation
* Infant aged up to 8 weeks

Exclusion Criteria:

* Do not speak French sufficiently well to participate in assessments
* Have established intellectual disability or psychotic illness
* Infant too instable regarding hemodynamic or respiratory functioning (severe brady apnea, more than 30% oxygen)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2016-08; Primary Completion 2020-02 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Perceived Maternal Parenting Self-Efficacy tool | 1 month

SECONDARY OUTCOMES:
Posttraumatic Diagnostic Scale | 1 month, 6 months
Parental Stressor Scale: Neonatal Intensive Care Unit | 1 month, 6 months
Parental Stress Index - Short form | 1 month, 6 months
Hospital Anxiety and Depression Scale | 1 month, 6 months
Edinburgh Postnatal Depression Scale | 1 month, 6 months
Mother-to-Infant Bonding Scale | 1 month, 6 months
Infant Behaviour Questionnaire - Revised very short form | 1 month, 6 months
Emotional Availability Scale | 6 months
Perceived Maternal Parental Self-Efficacy tool | 6 months
CARE-Index | 6 months

OTHER OUTCOMES:
Satisfaction with intervention questionnaire | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Antje Horsch, DClinPsych, Principal Investigator — Clinical and Research Psychologist
Locations (1):
- Neonatology Service, University Hospital Lausanne, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lovey O, Bickle-Graz M, Morisod Harari M, Horsch A, Schneider J; JOIN Research Consortium. The Joint Observation in Neonatology and Neurodevelopmental Outcome of Preterm Infants at Six Months Corrected Age: Secondary Outcome Data from a Randomised Controlled Trial. Children (Basel). 2022 Sep 13;9(9):1380. doi: 10.3390/children9091380. PMID 36138689
- [Derived] Schneider J, Borghini A, Morisod Harari M, Faure N, Tenthorey C, Le Berre A, Tolsa JF, Horsch A; JOIN Research Consortium. Joint observation in NICU (JOIN): study protocol of a clinical randomised controlled trial examining an early intervention during preterm care. BMJ Open. 2019 Mar 30;9(3):e026484. doi: 10.1136/bmjopen-2018-026484. PMID 30928952